CLINICAL TRIAL: NCT03781830
Title: A Pilot Study of Mobile Directly Observed Therapy (mDOT) for Immunosuppressant Adherence in Adolescent Liver Transplant Recipients
Brief Title: mDOT for Immunosuppressant Adherence in Adolescent Liver Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting under the new mDOT clinical trial with PI D Mogul
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00177456
Record Dates: First submitted 2018-06-07; First posted 2018-12-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Medication Adherence; Liver Transplantation
Keywords: mHealth; liver transplantation; medication adherence; video directly observed therapy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a single center prospective trial. Participants in this study will use the mHealth application to manage and track their immunosuppression medical regimen post-transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth Intervention (Experimental): Participants will receive the mHealth application either while they are an inpatient post-transplant, or at one of their post-transplant clinic visits. Study personnel will assist participants with downloading the mHealth application and explain its functioning. Participants will then use the application to aid in immunosuppressive medication adherence post-transplant.
  Interventions: Other: mHealth Intervention

INTERVENTIONS:
Other: mHealth Intervention — The video DOT app will allow transplant recipients to see their medication regimen, record themselves taking every dose, report side effects or symptoms, visualize their treatment progress, access educational content, and track appointments. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review.

SUMMARY:
The investigators are interested in whether or not the use of a mobile health (mHealth) application increases the rate of immunosuppression medication adherence among adolescent liver transplant recipients. The investigators aim to test this by recruiting adolescent (ages 14-21) liver transplant recipients to use an mHealth application to record themselves taking their immunosuppression medications, and tracking medication adherence over time. The study population will be approximately 25 adolescent liver transplant recipients at the Johns Hopkins Hospital.

DETAILED DESCRIPTION:
Non-adherence to immunosuppressive medications among organ transplant recipients is associated with a range of short- and long-term complications, and non-adherence is almost 4 times higher in pediatric and adolescent patients compared to adult transplant recipients. Previous studies have reported rates of non-adherence in this population ranging from 50-70%. Medication non-adherence in adolescents is associated with increased disease frustration, poor regimen adaptation/cognitive issues, difficulty with ingestion (e.g., number of medications, taste), and lack of parental monitoring and involvement. Among pediatric transplant recipients, psychosocial variables (e.g., psychiatric co-morbidities; child responsibility for medication) are strong determinants of nonadherence. Medication adherence is a key concern in the transition from pediatric to adult-centered transplant care, and transition planning should be prioritized in these transplant patients. Therefore, the investigators believe that the use of mobile health (mHealth) technology has the potential to allow clinicians and researchers to better understand nonadherence in pediatric transplant recipients, and increase immunosuppressive medication adherence.

The investigators will use a mobile health platform that enables users to track dose-by-dose medication adherence through asynchronous, video directly observed therapy (DOT). This helps patients take their medication as prescribed and gives providers the assurance that their patients are supported and successful in treatment. DOT is the practice of watching a patient take every dose of medicine in-person, and has typically only been done in extreme cases because it can be both costly and burdensome: DOT is the standard of care for Tuberculosis treatment and has proven high-adherence rates. Through mHealth technology, DOT can be used more broadly and without added burden; emocha's technology allows this through enabling patients to use their mobile application to view their regimen, record themselves taking every dose of their medication, report side effects or symptoms, visualize their treatment progress, and access educational content. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review. The aim of this study is to understand medication adherence in adolescent liver transplant recipients using the mHealth application.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (14-21 years old)
* Have received a liver transplant at the Johns Hopkins Hospital

Exclusion Criteria:

* Non-English speaking
* International

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
12-week immunosuppression adherence | 12 weeks
  After 12 weeks in the study, patients will complete the 4-item immunosuppressant therapy adherence instrument (ITAS) to determine self-reported medication adherence (scores range from 0-12 with 0 indicating very poor adherence and 12 indicating perfect adherence). Additionally, immunosuppression level trends will be tracked via electronic medical record review to determine medication adherence.

SECONDARY OUTCOMES:
Feasibility of using the mHealth Application as Assessed by a Semi-Structured Interview and a 17-Item Survey | 12 weeks
  After 12 weeks in the study, participants will be asked to participate in a semi-structured phone interview in which they will answer questions regarding their medication adherence habits and their thoughts on how our mHealth technology was or was not helpful. They will also complete a 17-question post-satisfaction survey assessing their satisfaction levels with the mhealth technology. Responses in the 17-item survey are on a 7-item Likert scale, ranging from Strongly Agree to Strongly Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Macey Henderson, JD, Phd, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Geest S, Borgermans L, Gemoets H, Abraham I, Vlaminck H, Evers G, Vanrenterghem Y. Incidence, determinants, and consequences of subclinical noncompliance with immunosuppressive therapy in renal transplant recipients. Transplantation. 1995 Feb 15;59(3):340-7. PMID 7871562
- [Background] Butler JA, Roderick P, Mullee M, Mason JC, Peveler RC. Frequency and impact of nonadherence to immunosuppressants after renal transplantation: a systematic review. Transplantation. 2004 Mar 15;77(5):769-76. doi: 10.1097/01.tp.0000110408.83054.88. PMID 15021846
- [Background] Foster BJ, Dahhou M, Zhang X, Platt RW, Samuel SM, Hanley JA. Association between age and graft failure rates in young kidney transplant recipients. Transplantation. 2011 Dec 15;92(11):1237-43. doi: 10.1097/TP.0b013e31823411d7. PMID 22124283
- [Background] Douglas S, Blixen C, Bartucci MR. Relationship between pretransplant noncompliance and posttransplant outcomes in renal transplant recipients. J Transpl Coord. 1996 Jun;6(2):53-8. doi: 10.7182/prtr.1.6.2.x11r325882657x21. PMID 9188358
- [Background] Burra P, Germani G, Gnoato F, Lazzaro S, Russo FP, Cillo U, Senzolo M. Adherence in liver transplant recipients. Liver Transpl. 2011 Jul;17(7):760-70. doi: 10.1002/lt.22294. PMID 21384527
- [Background] Mehta P, Steinberg EA, Kelly SL, Buchanan C, Rawlinson AR. Medication adherence among adolescent solid-organ transplant recipients: A survey of healthcare providers. Pediatr Transplant. 2017 Nov;21(7). doi: 10.1111/petr.13018. Epub 2017 Jul 2. PMID 28670855
- [Background] Dobbels F, Van Damme-Lombaert R, Vanhaecke J, De Geest S. Growing pains: non-adherence with the immunosuppressive regimen in adolescent transplant recipients. Pediatr Transplant. 2005 Jun;9(3):381-90. doi: 10.1111/j.1399-3046.2005.00356.x. PMID 15910397
- [Background] Fredericks EM, Lopez MJ, Magee JC, Shieck V, Opipari-Arrigan L. Psychological functioning, nonadherence and health outcomes after pediatric liver transplantation. Am J Transplant. 2007 Aug;7(8):1974-83. doi: 10.1111/j.1600-6143.2007.01878.x. PMID 17617862
- [Background] Pai AL, McGrady M. Systematic review and meta-analysis of psychological interventions to promote treatment adherence in children, adolescents, and young adults with chronic illness. J Pediatr Psychol. 2014 Sep;39(8):918-31. doi: 10.1093/jpepsy/jsu038. Epub 2014 Jun 20. PMID 24952359
- [Background] Shaw RJ, Palmer L, Blasey C, Sarwal M. A typology of non-adherence in pediatric renal transplant recipients. Pediatr Transplant. 2003 Dec;7(6):489-93. doi: 10.1046/j.1397-3142.2003.00117.x. PMID 14870900
- [Background] Simons LE, Blount RL. Identifying barriers to medication adherence in adolescent transplant recipients. J Pediatr Psychol. 2007 Aug;32(7):831-44. doi: 10.1093/jpepsy/jsm030. Epub 2007 May 23. PMID 17522111
- [Background] Simons LE, McCormick ML, Devine K, Blount RL. Medication barriers predict adolescent transplant recipients' adherence and clinical outcomes at 18-month follow-up. J Pediatr Psychol. 2010 Oct;35(9):1038-48. doi: 10.1093/jpepsy/jsq025. Epub 2010 Apr 20. PMID 20410021
- [Background] Kahana SY, Frazier TW, Drotar D. Preliminary quantitative investigation of predictors of treatment non-adherence in pediatric transplantation: a brief report. Pediatr Transplant. 2008 Sep;12(6):656-60. doi: 10.1111/j.1399-3046.2007.00864.x. PMID 18798360
- [Background] Berquist RK, Berquist WE, Esquivel CO, Cox KL, Wayman KI, Litt IF. Adolescent non-adherence: prevalence and consequences in liver transplant recipients. Pediatr Transplant. 2006 May;10(3):304-10. doi: 10.1111/j.1399-3046.2005.00451.x. PMID 16677353
- [Background] Watson AR. Non-compliance and transfer from paediatric to adult transplant unit. Pediatr Nephrol. 2000 Jun;14(6):469-72. doi: 10.1007/s004670050794. PMID 10872185
- [Background] Dobbels F, Ruppar T, De Geest S, Decorte A, Van Damme-Lombaerts R, Fine RN. Adherence to the immunosuppressive regimen in pediatric kidney transplant recipients: a systematic review. Pediatr Transplant. 2010 Aug;14(5):603-13. doi: 10.1111/j.1399-3046.2010.01299.x. Epub 2010 Feb 28. PMID 20214741
- [Background] Annunziato RA, Emre S, Shneider B, Barton C, Dugan CA, Shemesh E. Adherence and medical outcomes in pediatric liver transplant recipients who transition to adult services. Pediatr Transplant. 2007 Sep;11(6):608-14. doi: 10.1111/j.1399-3046.2007.00689.x. PMID 17663682
- [Background] Fredericks EM, Dore-Stites D, Well A, Magee JC, Freed GL, Shieck V, James Lopez M. Assessment of transition readiness skills and adherence in pediatric liver transplant recipients. Pediatr Transplant. 2010 Dec;14(8):944-53. doi: 10.1111/j.1399-3046.2010.01349.x. PMID 20598086
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):e147-e195. doi: 10.1093/cid/ciw376. Epub 2016 Aug 10. PMID 27516382
- [Background] Chisholm MA, Lance CE, Williamson GM, Mulloy LL. Development and validation of the immunosuppressant therapy adherence instrument (ITAS). Patient Educ Couns. 2005 Oct;59(1):13-20. doi: 10.1016/j.pec.2004.09.003. PMID 16198214